CLINICAL TRIAL: NCT04999228
Title: First-line Treatment With Infliximab Versus Corticosteroids in Children With Newly Diagnosed Moderate to Severe Ulcerative Colitis
Brief Title: Top Down Versus Step up in Pediatric Ulcerative Colitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Ying HUANG, Chief of Gastroenterology, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UC1.1
Record Dates: First submitted 2021-08-05; First posted 2021-08-10 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Ulcerative Colitis; Infliximab; Children
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Infliximab; Mesalamine; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infliximab treatment group (Experimental): For newly diagnosed moderate to severe Pediatric ulcerative colitis, infliximab will be used as first-line treatment
  Interventions: Drug: Infliximab
- Corticosteroid treatment group (Active Comparator): For newly diagnosed moderate to severe Pediatric ulcerative colitis, corticosteroids will be used as first-line treatment
  Interventions: Drug: Corticosteroids

INTERVENTIONS:
Drug: Infliximab — Infliximab will be administered intravenously at a dose of 5 mg/kg for 0, 2, and 6 weeks, then every 8 weeks for 1 year.
  Other Names: 5-ASA, AZA
  Arms: Infliximab treatment group
Drug: Corticosteroids — Corticosteroid will be given at a dose of 1-2mg/kg/day (maximum 60 mg/kg/day),oral or intravenously for 12 to 14 weeks.
  Other Names: 5-ASA, AZA
  Arms: Corticosteroid treatment group

SUMMARY:
Pediatric Ulcerative Colitis (UC) patients with moderate to severe disease activity at high risk of colectomy. Early use of biologic agents will likely be more effective. But there were no studies identified that compared a strategy of upfront biologic-based therapy versus gradual step-up therapy. In our study, newly diagnosed moderate to severe pediatric UC patients (6-18 years old) will be randomly divided into infliximab (IFX) treatment group (Top down group, TD) and corticosteroids (CS) treatment group (Step-up group, SU). Mucosal healing rate at week 12 will be compared between the two groups. The relapse rates and sustained durations of remission within one year will also be evaluated.

DETAILED DESCRIPTION:
Pediatric ulcerative colitis (UC) is typically more extensive and has a more active disease course than adult UC. Pediatric UC patients with moderate to severe disease activity at high risk of colectomy. Rapid disease control may improve the prognosis of the disease and reduce the rate of surgery. Early use of biologic agents will likely be more effective. But there were no studies identified that compared a strategy of upfront biologic-based therapy versus gradual step-up therapy. In our study, newly diagnosed moderate to severe pediatric UC patients (6-18 years old) will be randomly divided into infliximab (IFX) treatment group (Top down group, TD) and corticosteroids (CS) treatment group (Step-up group, SU). A decrease of pediatric ulcerative colitis activity index (PUCAI) at least 20 points were defined as Clinical response. Clinical response will be evaluated at week 2 in SU group and week 6 in TD group. For no-responder, treatment plan will be changed. Clinical remission rate at week 10 and mucosal healing rate at week 12 will be compared between the two groups. The relapse rates and sustained durations of remission within one year will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. newly diagnosed UC;
2. moderate to severe disease activity
3. Age: 6 to 18 years old

Exclusion Criteria:

1. with mild disease activity
2. Have been treated with Corticosteroid or biological agents for UC

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mucosal healing rate | 12 week after intervention
  The Ulcerative Colitis Endoscopic Index of Severity (UCEIS) ≦1 points is defined as mucosal healing. This will be evaluated by inflammatory bowel disease endoscopist.

SECONDARY OUTCOMES:
The relapse rates | 1 year after intervention
  Relapse is defined as an increased in pediatric Ulcerative Colitis activity index (PUCAI) score by 10 points or more after clinical remission or when new Ulcerative Colitis treatment needed to be started due to worsening of symptoms. This will be evaluated by gastroenterologist.
Sustained durations of remission | 1 year after intervention
  Sustained pediatric Ulcerative Colitis activity index (PUCAI) score <10 points during follow-up（week 10 to week 54 after intervention). This will be evaluated by gastroenterologist.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Huang, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China